CLINICAL TRIAL: NCT02696707
Title: An Integrated Consent Model Study to Compare Two Standard of Care Schedules for Monitoring Cardiac Function in Patients Receiving Trastuzumab for Early Stage Breast Cancer
Acronym: OTT 15-05
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20150777-01H
Record Dates: First submitted 2016-02-18; First posted 2016-03-02 (Estimated); Results first posted 2025-07-14 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: cardiac toxicities
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LVEF 3 month (Active Comparator): cardiac evaluation (by either transthoracic echocardiography or MUGA) every 3 months
  Interventions: Procedure: LVEF 3 month
- LVEF 4 month (Active Comparator): cardiac evaluation (by either transthoracic echocardiography or MUGA) every 4 months
  Interventions: Procedure: LVEF 4 month

INTERVENTIONS:
Procedure: LVEF 3 month — cardiac evaluation (by either transthoracic echocardiography or MUGA) every 3 months
  Arms: LVEF 3 month
Procedure: LVEF 4 month — cardiac evaluation (by either transthoracic echocardiography or MUGA) every 4 months
  Arms: LVEF 4 month

SUMMARY:
Several large adjuvant trastuzumab trials have demonstrated improved overall survival in participants with early stage breast cancer, with a 33% decrease in risk of death. However, retrospective analyses of participant outcomes in these trials have demonstrated increased risk of cardiotoxicity (i.e damage to the heart) in a small number of patients (4-8%).

At this time, investigators are unable to predict which participants are at increased risk of cardiac-related treatment complications. Currently all patients receive regular cardiac imaging throughout their one year of trastuzumab treatment.

At this time, the optimal monitoring schedule for trastuzumab-related cardiotoxicity remains unknown, and several published consensus guidelines are currently in use as standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed early stage HER2-positive breast cancer
* Planned trastuzumab therapy for early stage breast cancer
* ≥18 years of age
* Able to provide verbal consent
* Normal LVEF (>53%) before trastuzumab therapy

Exclusion Criteria:

• Contraindication to transthoracic echocardiography or MUGA

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-06; Primary Completion 2020-05 (Actual); Study Completion 2020-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olexiy Aseyey, MD, Principal Investigator — The Ottawa Hospital
Locations (4):
- Canada (4):
  - Southlake Regional Health Centre, Newmarket, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dent S, Fergusson D, Aseyev O, Stober C, Pond G, Awan AA, McGee SF, Ng TL, Simos D, Vandermeer L, Saunders D, Hilton JF, Hutton B, Clemons M. A Randomized Trial Comparing 3- versus 4-Monthly Cardiac Monitoring in Patients Receiving Trastuzumab-Based Chemotherapy for Early Breast Cancer. Curr Oncol. 2021 Dec 3;28(6):5073-5083. doi: 10.3390/curroncol28060427. PMID 34940066
- See also: Rethinking Clinical Trials (REaCT) Website — https://react.ohri.ca/

RESULTS

PARTICIPANT FLOW:
Period: Per Protocol Population
Arm/Group | LVEF 3 Month | LVEF 4 Month
Started | 100 | 100
Completed | 98 | 97
Not Completed | 2 | 3
Not completed — Physician Decision | 2 | 1
Not completed — Participant Decision | 0 | 2
Period: Completed Study as Planned
Arm/Group | LVEF 3 Month | LVEF 4 Month
Started | 98 | 97
Completed | 90 | 88
Not Completed | 8 | 9
Not completed — Reason = LVEF | 2 | 2
Not completed — Protocol Violation | 2 | 6
Not completed — Metastatic disease | 3 | 0
Not completed — Location | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LVEF 3 Month | LVEF 4 Month | Total
Number analyzed (Participants) | 98 | 97 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (11.4) | 54.8 (11.3) | 55.1 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 97 | 195
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Baseline Left Ventricular Ejection Fraction (LVEF) [Median (Full Range); unit: LVEF Percentage (%)] — Baseline LVEF measured by echocardiogram or MUGA and reported as a percentage
  LVEF Percentage (%) | 65 [54 to 82] | 64 [54 to 76] | 65 [54 to 82]
Anthracycline-based chemotherapy [Count of Participants; unit: Participants] | 53 | 50 | 103

OUTCOME MEASURES:

1. Primary Outcome: LVEF Results
Description: Changes in Left Ventricular Ejection Fraction (LVEF) results compared to baseline (by echocardiography or MUGA) throughout the course of trastuzumab based therapy. LVEF is measured as a percentage. The outcome is a change in LVEF percentage (%).
Time Frame: Baseline to 1 year
Population: Per Protocol Population
Measure: Median (Full Range); unit: LVEF Percentage (%)
Arm/Group | LVEF 3 Month | LVEF 4 Month
Number analyzed (Participants) | 98 | 97
LVEF Percentage (%) | -8 [-26 to 17] | -6 [-33 to 10]
Statistical Analysis 1: Comparison: LVEF 3 Month vs LVEF 4 Month; Test type: Non-Inferiority — The non-inferiority margin between groups was set as 4%; Difference = -0.6, 95% CI 2-sided [-2.5 to 1.2]

2. Secondary Outcome: Rates of Trastuzumab Delay and Discontinuation
Description: The number of participants who had a delay and/or discontinuation in trastuzumab treatment. Data was collected from physicians following clinic visits and from patient electronic medical records.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | LVEF 3 Month | LVEF 4 Month
Number analyzed (Participants) | 98 | 97
Participants
  Delay | 9 | 2
  Discontinuation | 2 | 7

3. Secondary Outcome: Referral to Cardiology
Description: The number of participants who were referred to cardiology. Data was collected from physicians following clinic visits, and from the patient's electronic medical record.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | LVEF 3 Month | LVEF 4 Month
Number analyzed (Participants) | 98 | 97
Participants | 12 | 12

4. Secondary Outcome: Rate of Cardiac Events
Description: The number of participants who experienced a decrease in ejection fraction (EF), congestive heart failure, or other cardiac events within the 1 year of study. Examples of other cardiac events include change in blood pressure, chest pain/shortness of breath, or irregular heartbeat. Data was collected/reported from physicians following clinic appointments, and from the patient's electronic medical record.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | LVEF 3 Month | LVEF 4 Month
Number analyzed (Participants) | 98 | 97
Participants | 31 | 24

ADVERSE EVENTS:
Time Frame: All-cause mortality was monitored for 12 months.
Description: Serious adverse event reporting was not required for this study, as per the protocol. This was a pragmatic clinical trial comparing two standard of care schedules of cardiac monitoring, not treatments. Cardiac adverse events were collected and reported as secondary clinical outcomes. They were not collected/reported as adverse events.
Arm/Group | LVEF 3 Month | LVEF 4 Month
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/97
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-13): https://cdn.clinicaltrials.gov/large-docs/07/NCT02696707/Prot_SAP_000.pdf